CLINICAL TRIAL: NCT01896791
Title: Transcranial Direct Current Stimulation (tDCS) in Vasomotor Symptoms of Menopause: Blind Sham Controlled Randomized Clinical Trial
Brief Title: Transcranial Direct Current Stimulation (tDCS) in Vasomotor Symptoms of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-0418
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Active Comparator): Active Transcranial Direct Current Stimulation: the anode electrode is placed in the area of the motor cortex M1 C3 or C4 position of the dominant hemisphere (International 10-20 EEG System). The cathode electrode is placed over the contralateral supraorbital region to the anode electrode. Treatment time and intensity of the stimulus: tDCS: 2mili Ampere, 20min, 10 days.
  Interventions: Procedure: Transcranial Direct Current Stimulation
- Sham Stimulation (Placebo Comparator): Sham Stimulation: appliance off during the entire period without active stimulation, with the position of the electrodes in the same sites of active stimulation
  Interventions: Procedure: Sham Stimulation

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation — Active Transcranial Direct Current Stimulation : the anode electrode is placed in the area of the motor cortex M1 C3 or C4 position of the dominant hemisphere (International 10-20 EEG System). The cathode electrode is placed over the contralateral supraorbital region to the anode electrode. Treatment time and intensity of the stimulus: tDCS: 2 mili Ampere, 20min, 10 days.
  Arms: Transcranial Direct Current Stimulation
Procedure: Sham Stimulation — Sham Stimulation- appliance off during the entire period without active stimulation, with the position of the electrodes in the same sites of active stimulation
  Arms: Sham Stimulation

SUMMARY:
Climacteric or Menopausal Transition is defined as the time period where there is a change to non-reproductive reproductive life, with extension of variable length. During this period, and after the establishment of Menopause and non-functioning ovarian, the appearance of various symptoms that express the depletion of ovarian follicles is common; among these symptoms, the most frequently reported by women are vasomotor symptoms or hot flashes. In addition to hormonal therapy, other medications have been employed in an attempt to improve these symptoms; although they present better results than placebo, yet have little clinical impact in reducing vasomotor symptoms. Therefore, this gap allows the evaluation of alternative therapies, such as Transcranial Direct Current Stimulation (tDCS). The rationale for studying the effect of this technique in this context is its possible autonomic modulatory effect. What reinforces the choice of this technique is the fact that it demonstrated efficacy in other pathologies such as depression, pain, Parkinson's disease, among others. Transcranial direct current stimulation (tDCS) is a renewed method of non-invasive brain modulation. It is based on a transcranial application of weak direct currents in a non-invasive, simple and painless manner. Its use in the treatment of vasomotor symptoms has not been studied. The objective of this study is to evaluate the improvement of vasomotor symptoms in postmenopausal women, after application of tDCS, and compare them to a control group. This Randomized Clinical Trial will be held in female postmenopausal patients, followed in the outpatient Menopause Clinic of Obstetrics and Gynecology Service, Hospital de Clinicas de Porto Alegre. From these results, it is expected to present a new therapeutic option in the treatment of vasomotor symptoms.

DETAILED DESCRIPTION:
Primary Outcome: evaluate the effect of tDCS on vasomotor symptoms in postmenopausal women treated at a tertiary hospital in southern Brazil.

Secondary Outcome: compare the effect of tDCS with sham-tDCS in postmenopausal women on vasomotor symptoms, FSH (Follicle Stimulating Hormone) levels, salivary cortisol, BDNF (Brains derived neurotrophic factor)levels,depressive symptoms and quality of life.

Interventions:

* Application of tDCS for a period of 10 consecutive days.
* Transcranial direct current stimulation (tDCS):

Active stimulation: the anode electrode is placed in the area of the motor cortex M1 C3 or C4 position of the dominant hemisphere (International 10-20 EEG System). The cathode electrode is placed over the contralateral supraorbital region to the anode electrode. Treatment time and intensity of the stimulus: 2 mili Ampere, 20min, 10 days.

Placebo-sham: appliance off during the entire period without active stimulation, with the position of the electrodes in the same sites of active stimulation.

The placebo group do not receive pharmacological treatment or other during the research.

After treatment, patients will be reassessed in a week, a month and three months with new application of questionnaires and sample collection.

ELIGIBILITY:
Inclusion Criteria:

menopause women, any age, with at least, eight hot flashes/day

Exclusion Criteria:

neurological or psychiatric diseases, patients with head injury, women in hormonal replacement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
number of diary vasomotor symptoms | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Maria Celeste Wender, PhD, Principal Investigator — Hospítal de Clinicas de Professor
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided